CLINICAL TRIAL: NCT05369052
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Contezolid Acefosamil and Contezolid Compared to Linezolid Administered Intravenously and Orally to Adults With Moderate or Severe Diabetic Foot Infections (DFI)
Brief Title: Safety and Efficacy Study of Contezolid Acefosamil and Contezolid Compared to Linezolid Administered Intravenously and Orally to Adults With Moderate or Severe Diabetic Foot Infections (DFI)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MicuRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRXC-302
Record Dates: First submitted 2022-04-12; First posted 2022-05-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Infection
MeSH Terms: interventions — Linezolid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- contezolid acefosamil/contezolid (Experimental)
  Interventions: Drug: contezolid acefosamil (IV)/contezolid (PO)
- linezolid (Active Comparator)
  Interventions: Drug: Linezolid (IV and PO)

INTERVENTIONS:
Drug: contezolid acefosamil (IV)/contezolid (PO) — Contezolid acefosamil (IV)/contezolid (PO) administered for a total of 14 to 28 days (28 to 56 doses)
  Arms: contezolid acefosamil/contezolid
Drug: Linezolid (IV and PO) — Linezolid (IV and PO) administered for a total of 14 to 28 days (28 to 56 doses)
  Arms: linezolid

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, safety and efficacy study of contezolid acefosamil (IV)/contezolid (PO) compared with linezolid (IV and PO) administered for a total of 14 to 28 days in adult subjects with moderate or severe DFI.

DETAILED DESCRIPTION:
Approximately 865 subjects (519 contezolid acefosamil/contezolid: 346 linezolid) will be enrolled with moderate or severe DFI that are confirmed or suspected to be due to a Gram-positive bacterial pathogen (MITT analysis set).

ELIGIBILITY:
Inclusion Criteria:

* Have diabetes mellitus (type 1 or 2) per the American Diabetes Association criteria
* Have a foot infection that started at or below the malleolus and does not extend above the knee
* Foot infection that meets the IWGDF DFI criteria for classification 3 (moderate infection) or 4 (severe infection)
* Foot infection had acute onset or worsening of signs and symptoms within the past 14 days

Exclusion Criteria:

* Previous DFI known or suspected to be caused by Gram-positive pathogens that are resistant to oxazolidinone antibiotics
* DFI with presumptive evidence or suspicion of osteomyelitis
* Necrotizing fasciitis, crepitant cellulitis, wet gangrene, gas gangrene, ecthyma gangrenosum, septic arthritis, or severely impaired arterial supply to any portion of the affected foot which may need revascularization before the end of the study
* Evidence of significant hepatic, renal, hematologic, or immunologic disease
* Females who are pregnant or breastfeeding
* Prior receipt of any formulation of contezolid acefosamil or contezolid
* Inability to cooperate fully with the requirements of the study protocol, including the schedule of events, or likely to be noncompliant with any study requirements, or the Investigator determines that the subject should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response calculated with percentage of subjects with resolution of DFI signs and symptoms and requiring no further therapy as assessed by Investigators | Day 35
  The primary objective is to evaluate the Investigator's assessment of clinical response at the D35 visit in subjects receiving contezolid acefosamil/contezolid compared to subjects receiving linezolid in the MITT analysis
Adverse events - symptoms reported by subjects | 28-35 days after End-of-Therapy (EOT)
  Evaluate safety of contezolid acefosamil (IV)/contezolid (PO) compared with linezolid (IV and PO)
Clinical laboratory assessment - complete blood count | 28-35 days after End-of-Therapy (EOT)
  Will be evaluated under safety of contezolid acefosamil (IV)/contezolid (PO) compared with linezolid (IV and PO)
Vital signs - heart rate | 28-35 days after End-of-Therapy (EOT)
  Will be evaluated under safety of contezolid acefosamil (IV)/contezolid (PO) compared with linezolid (IV and PO)

SECONDARY OUTCOMES:
Clinical response calculated with percentage of subjects with resolution of DFI signs and symptoms and requiring no further therapy as assessed by Investigators | 14-28 days
  Evaluate the Investigator's assessment of clinical response at EOT visit in the MITT analysis set
Clinical response calculated with percentage of subjects with resolution of DFI signs and symptoms and requiring no further therapy as assessed by Investigators | Day 10, 28-35 days after EOT
  Evaluate the Investigator's assessment of clinical response at Day 10 (D10) and Late Follow-Up visits (LFU; 28-35 days after EOT) in the MITT analysis set

CONTACTS AND LOCATIONS:
Locations (14):
- United States (2):
  - New Hope Research Development, Corona, California
  - ILD Research Center, Vista, California
- Bulgaria (4):
  - MHAT Sveti Nikolay Chudotvorets EOOD, Lom
  - Multiprofile Hospital for Active Treatment - KANEV, Rousse
  - Medical Institute Ministry of Interior Central Clinical Base, Sofia
  - University Multidisciplinary Hospital for Active Treatment and Emergency Medicine 'N. I. Priogov´, Sofia
- South-Estonian Hospital Ltd., Võru, Estonia
- Georgia (2):
  - LTD High Technology Hospital Med Center, Batumi
  - JSC Vian - West Georgia Medical Center, Kutaisi
- GMV Care& Research - Maria Cecilia Hospital, Cotignola, Italy
- Daugavpils Regional Hospital, Daugavpils, Latvia
- Poland (2):
  - Instytut Medycyny Wsi im. W. Chodzki, Lublin
  - PODEMA Sp. z o.o., Warsaw
- University Clinical Center Kragujevac, Kragujevac, Serbia

IPD SHARING:
Plan to Share IPD: No